CLINICAL TRIAL: NCT04178499
Title: Smoking: Cytokines in Vitreous and Aqueous Humor
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 30-107 ex 17/18
Record Dates: First submitted 2019-11-18; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Vitreous humor Aqueous humor Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smokers: active smokers
  Interventions: Diagnostic Test: cytokine analysis
- non-smokers: never smokers
  Interventions: Diagnostic Test: cytokine analysis

INTERVENTIONS:
Diagnostic Test: cytokine analysis — analysis of intraocular cytokines

SUMMARY:
Smoking is a risk factor for ophthalmologic diseases. Inflammation might play a role in their pathogenesis.

This study elucidates intraocular cytokine profiles in smokers and non smokers.

ELIGIBILITY:
Inclusion Criteria:

* scheduled vitrectomy and/or cataract surgery
* signed informed consent

Exclusion Criteria:

* diabetes
* uveitis
* rheumatologic disease
* anti-inflammatory/immunomodulatory medications
* st.p. intravitreal injections
* st.p. glaucoma surgery
* cataract surgery on the eye to be examined within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for vitrectomy at the Medical University of Graz/Austria
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
cotinine | At the time of vitrectomy procedure
  Concentration of intraocular cotinine

IPD SHARING:
Plan to Share IPD: No